CLINICAL TRIAL: NCT04680169
Title: I-gel Versus AuraGain for Bronchoscopic Intubation Through Supraglottic Airway Device - a Randomized Controlled Trial
Brief Title: I-gel vs AuraGain for Bronchoscopic Intubation Through SGA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Intubation through SGA
Record Dates: First submitted 2020-12-17; First posted 2020-12-22 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2020-12

CONDITIONS: Airway Management
Keywords: Intubation; Bronchoscopic; Supraglottic airway device; I-gel; AuraGain; Flexible; Fiberoptic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Bronchoscopic intubation using AuraGain LMA as conduit (Active Comparator): A group of 50 patients randomly allocated to bronchoscopic intubation using AuraGain
  Interventions: Device: Bronchoscopic intubation through AuraGain LMA
- Group B: Bronchoscopic intubation with I-gel SGA as conduit (Active Comparator): A group of 50 patients randomly allocated to bronchoscopic intubation using I-gel
  Interventions: Device: Bronchoscopic intubation through I-gel SGA

INTERVENTIONS:
Device: Bronchoscopic intubation through AuraGain LMA — Comparing two different SGAs as conduit for bronchoscopic tracheal intubation
  Arms: Group A: Bronchoscopic intubation using AuraGain LMA as conduit
Device: Bronchoscopic intubation through I-gel SGA — Comparing two different SGAs as conduit for bronchoscopic tracheal intubation
  Arms: Group B: Bronchoscopic intubation with I-gel SGA as conduit

SUMMARY:
This trial compares two different second generation supraglottic airway devices (AuraGain and I-gel) used as a conduit for bronchoscopic tracheal intubation during continuous oxygenation in order tο determine time to successful tracheal intubation and ease of use.

DETAILED DESCRIPTION:
A prospective randomized controlled trial in the Department of Anesthesiology, Copenhagen University Hospital Nordsjællands Hospital-Hillerød Denmark. The study is approved by the Ethics Committee, capital region of Denmark. The aim of the study is to compare bronchoscopic tracheal intubation during continuous oxygenation through the AuraGain and I-gel supraglottic airway device. One hundred patients will be randomly allocated into two groups, group A (AuraGain) and group B (I-gel). Study outcomes are time to tracheal intubation confirmed by capnography as well as anesthesiologists reports of ease of use. Twenty-five anesthesiologists participates in this study, and are allocated four patient each. In random order, each physician will perform two bronchoscopic tracheal intubations with each SGA.

In the preoperative setting, a complete anesthetic evaluation will be performed, including a detailed airway assessment determining predictors for difficulties of face mask ventilation, insertion of SGA and tracheal intubation. Participants are scheduled to undergo elective surgery under general anesthesia. Before induction, all patients will be preoxygenated with 100% oxygen. After induction, rocuronium 0.6mg/kg will be used to facilitate neuromuscular blockade. Sufficient face mask ventilation will be performed before intervention.

Group A: AuraGain:

Time is measured from when the anesthesiologist reaches for the AuraGain LMA until the mask is placed and adequate ventilation is confirmed by capnography. The AuraGain LMA will be used as conduit for bronchoscopic intubation during continuous oxygenation, and time is measured until placement of the tracheal tube verified by capnography.

Group B: I-gel:

Time is measured from when the anesthesiologist reaches for the I-gel LMA until the mask is placed and adequate ventilation is confirmed by capnography.The I-gel LMA will be used as conduit for bronchoscopic tracheal intubation during continuous oxygenation, and time is measured until placement of the tracheal tube verified by capnography.

In both groups (A and B) up to two attempts of SGA placement and up to three attempts of tracheal intubation are allowed.

In case of an emerging unpredicted difficult airway and a concurrent unsuccessful SGA placement, the difficult airway algorithm, DAS, UK will be followed. Video- assisted laryngoscopy will be the first option.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for a non-acute ENT, gynaecological, gastrointestinal or orthopaedic surgical procedure for which general anaesthesia including oral intubation with an endotracheal tube will be provided

Exclusion Criteria:

* Age<18 years
* Inter-incisional distance <30mm
* Pregnant and BMI>40kg/m2
* ASA physical status classification system grade >3
* Earlier laryngeal or pharyngeal surgery
* Increased risk of aspiration (e.g. nasogastric tube inserted, planned Rapid Sequence Induction)
* Informed consent cannot be obtained
* Patients with stridor
* Patients with hypoxemia defines by saturation <90 without oxygen at arrival to the operating room
* Use of oxygen supply at home
* Need of one of the following special endotracheal tubes for scheduled surgery: neural integrity monitor (NIM) electromyogram (EMG) tracheal tubes, wire tubes
* Patients scheduled for any awake approach to secure the airway e.g. awake videolaryngoscopy, awake fiberoptic bronchoscope intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

PRIMARY OUTCOMES:
Total time for airway management | Up to study completion, an average of 4 months
  Total time from reaching the SGA with hands to ended bronchoscopic tracheal intubation confirmed by the end of first curve on capnography

SECONDARY OUTCOMES:
Time to placement of SGA | Up to study completion, an average of 4 months
  Time measured from reaching SGA with hands to correct placement of SGA confirmed by end of first curve on capnography
Time to trans-device tracheal intubation | Up to study completion, an average of 4 months
  time measured from confirmed placement of SGA until successful tracheal intubation confirmed by end of first curve on capnography
Number of attempts needed for correct placement of SGA | Up to study completion, an average of 4 months
  two attempts at correct placement allowed. Attempt is failed if no curve appears on capnography.
Number of attempts needed for correct intubation | Up to study completion, an average of 4 months
  Attempt of bronchoscopic intubation begins when entering aScope in swivel. Attempt is failed if airway is not visualised, if tracheal tube can not be advanced in trachea, if SpO2 is <85% or if total time exceeds 6 minutes. Three attempts of intubation is allowed.

OTHER OUTCOMES:
Reason for failed intubation | Up to study completion, an average of 4 months
  if failed (as described in outcome 4), reason of failure is described
Feeling of resistance during tracheal intubation | Up to study completion, an average of 4 months
  Physician will be asked to report resistance as: none, mild, severe, impossible
Feasibility of SGA placement | Up to study completion, an average of 4 months
  Physician will be asked to report feasibility at a scale 1-10, 1=easy, 10=very difficult
Feasibility of intubation | Up to study completion, an average of 4 months
  Physician will be asked to report feasibility at a scale 1-10, 1=easy, 10=very difficult
Feasibility of total airway management | Up to study completion, an average of 4 months
  Physician will be asked to report feasibility of the whole procedure at a scale 1-10, 1=easy, 10=very difficult
Best Brimacombe score | Up to study completion, an average of 4 months
  Class 1: Unable to see the vocal cords. Class 2: the vocal cords and the anterior aspect of the epiglottis are visualized. Class 3: the vocal cords and the posterior aspect of the epiglottis are observed. Grade 4: only vocal cords were observed.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte V Rosenstock, Ph.d, Principal Investigator — Nordsjaellands Hospital
Locations (1):
- Nordsjaellands Hospital, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: No